CLINICAL TRIAL: NCT04286139
Title: Self-management and HeAlth Promotion in Early-stage Dementia With E-learning for Carers - SHAPE: A Multicentre, Randomised, Controlled Trial
Brief Title: Self-management and HeAlth Promotion in Early-stage Dementia With E-learning for Carers
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: The Research Council of Norway (Other); Alzheimer's Society (Other); National Health and Medical Research Council, Australia (Other); University of Exeter (Other); London School of Economics and Political Science (Other); The University of New South Wales (Other); The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 258388
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2021-08

CONDITIONS: Dementia
Keywords: Health promotion; Self-management; Online
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHAPE Intervention (Experimental): This group will receive the online group based self-management course develop self-management skills in areas including decision making, symptom management and social interaction and to provide information on the disease process and the development of healthy behaviours in a supportive learning environment to prevent problems that are common in the later stages of the disease. Key themes of the intervention will include positive actions to improve and maintain health, how to talk about the impact of the disease on the life of the person with dementia, fear of losing independence and how to tackle and solve other sensitive issues. Running in parallel there will be an e-learning resource available to the carers which covers the similar material covered in the group sessions for the person with dementia, as well as some additional resources and signposting to help them in their role supporting the person with dementia.
  Interventions: Behavioral: SHAPE
- Treatment as usual (No Intervention): Participants in the TAU arm will receive normal services such as clinical reviews, psychiatric appointments and other services when needed. With TAU as the comparator condition ensures that participants receive any needed services and enable comparison between current best practice and the new intervention of SHAPE

INTERVENTIONS:
Behavioral: SHAPE — The SHAPE intervention provides information for carers, and maintains the dignity and autonomy of the person with dementia, supporting them in planning for the future with their family. The person with dementia attends an online 10 week facilitator lead group based course. It is designed to develop self-management skills in areas including decision-making, symptom management and social interaction. It also provides information on the disease process and the development of healthy behaviors in a supportive learning environment to prevent problems that are common in the later stages of the disease. The adjunctive e-learning platform for carers provides the same information that the person with dementia receives plus additional material and signposting to support them in their role. This will empower the whole family to support and enable more effective self-management by the person with dementia, and enhance their ability to plan ahead together and make key decisions jointly.
  Arms: SHAPE Intervention

SUMMARY:
This study aims to assess if an educational programme combining approaches of self-management, health promotion, and e-learning will improve self-efficacy and other key health and mental health outcomes for people with mild to moderate dementia.

DETAILED DESCRIPTION:
It is currently estimated that 47 million people are living with dementia today and this number is expected to double in the next 20 years. Unfortunately, there has been limited advancement in medical treatments for dementia and new cost-effective approaches are needed. The utility of self-management has been proven to be of benefit in certain chronic diseases, however, very little work has been undertaken regarding self-management in people with dementia.The SHAPE self-management group therapy aims to significantly improve self-efficacy in people with mild to moderate dementia and to improve key health and mental health outcomes, carer stress and knowledge of dementia.SHAPE comprises a 10 week online course delivered as group sessions for the participants with dementia. The sessions are designed to develop self-management skills and to provide information on the disease process and the development of healthy behaviours in a supportive learning environment to prevent problems that are common in the later stages of the disease. E-learning resources will be provided for carers (study supporters) which covers the similar and complimentary material discussed in the group sessions for the participant with dementia.

This trial uses 2:1 randomisation and will assess the clinical and cost effectiveness of SHAPE. Participants will be randomised to participate in the SHAPE intervention or continue with usual care. To assess the effectiveness of SHAPE at improving self-efficacy and secondary outcomes a battery of questionnaires will be administered to the participants and study supporters at baseline, after SHAPE participants have completed the intervention, and 9 months after randomisation. The answers to these questionnaires will be assessed and the results compared between the two groups of participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia according to the ICD-10 classification or the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV or V
* 65 years of age or older
* Mild to moderate dementia, as associated with tMMSE ≥15
* Ability to read and write
* Hearing and vision that are sufficiently good to work in a group setting
* Capacity to give consent for participation in the study
* Proficient in the language in which the intervention is provided
* Care partner willing to participate

Exclusion Criteria:

* A diagnosis of alcohol or drug abuse
* Lewy body dementias, Fronto-temporal lobar degeneration or Semantic dementia
* A limited life expectancy due to any terminal disease or other serious illness, other than dementia
* Chemotherapy or radiation treatment ongoing at enrolment
* Currently participating in health promotion or self-management group

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in general self-efficacy | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the General Self-Efficacy Scale, a 10-item psychometric scale where each item is scored on a 4 point scale ranging from 'Not at all true' to 'Hardly true', to assess optimistic self-beliefs to cope with a variety of difficult demands in life.

SECONDARY OUTCOMES:
Change in mood (anxiety, depression) | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Cornell Scale for Depression in Dementia (CSDD) for participants with dementia. Scale ranges from 0-38, where high score indicates high symptom load.
Change in wellbeing | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Sense of Competence Questionnaire Short version (SSCQ). This is a 7-item questionnaire, scale scores range from 7-35, where higher scores indicate higher sense of competence, which is an important factor in their wellbeing.
Change in Health-related Quality of life (HRQL) | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Dementia Quality of Life Scale (DEMQOL) for participants with dementia. A 28 item interviewer-administered questionnaire with a score range of 28 to 112, higher scores indicating better HRQL.
Change in Health-related Quality of life (HRQL) | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Dementia Quality of Life Scale (DEMQOL) proxy version. A 31 item interviewer-administered questionnaire answered by a carer with a score range of 31 to 124, higher scores indicating better HRQL.
Change in Quality of life | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by EQ-5D-5L. Descriptive measure of quality of life comprising 5 Dimensions With 5 Levels each, scores can be converted to a single summary index number. A visual analog scale records self-rated health ranging 0-100, high score indicates good health.
Change in health behaviours | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by Self-reported health behaviour change questionnaire. Comprises 17 questions about specific health-related change that occurred during each time period, and if yes, how much of a change ranging from 'a little change', 'quite a bit of change', and 'great change'.
Change in cognition | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the telephone Mini-Mental Status Examination (tMMSE). Assesses cognitive function in people with dementia. With a maximum score of 26, lower scores indicate greater cognitive issues.
Cognition and function | Baseline
  Measured by the Modified Clinical Dementia Rating Scale (mCDR), a 5-point likert scale used to characterize six domains of cognitive and functional performance, level of impairment/dementia is ranging from 0=Normal, 0.5 = Very Mild Dementia, 1 = Mild Dementia, 2 = Moderate Dementia, 3 = Severe Dementia
Change in function | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Functional Activities Questionnaire (FAQ). 10 items measuring instrumental activities of daily living (IADLs), with sum score ranging 0-30. Higher score indicates impaired function.
Change in neuropsychiatric symptoms | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Neuropsychiatric Inventory Questionnaire (NPI-Q), an informant based questionnaire assessing the presence and severity of 12 Neuropsychiatric Symptoms. Severity scores range from 0-36, where higher scores indicate more severe behavioural and psychological symptoms of dementia. Distress scores range from 0-60, where higher values represent higher levels of distress due to symptoms.
Change in carer stress | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Relative Stress Scale (RSS), which consists of 15 items ranging from 0-4, high score indicates high burden on carers.
Change in knowledge about dementia | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Dementia Knowledge Assessment Scale (DKAS). Comprising 25 items with statements about the condition, including general characteristics, symptoms, risk factors, care and treatment. Respondents answer on a modified Likert scale with five response options: false, probably false, probably true, true, don't know.
Change in perceived access to service use | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Client Service Receipt Inventory (CSRI). A validated tool to gather information on current living arrangements, medication, use of hospital, community-based and day services.
Change in cost of care | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by the Client Service Receipt Inventory (CSRI). A validated tool to gather information on current living arrangements, medication, use of hospital, community-based and day services.
Change in quality of adjusted life-years (QALY) | Baseline to 3 months (primary time-point), and 9 months after baseline (follow-up)
  Measured by EuroQoL Instrument EQ-5D-5L. Descriptive measure of quality of life comprising 5 Dimensions With 5 Levels each, scores can be converted to a single summary index number. A visual analog scale records self-rated health ranging 0-100, high score indicates good health.

OTHER OUTCOMES:
Promoting and hindering factors of the intervention | 3 months (Primary time-point)
  Measured using post-intervention qualitative interviews with intervention facilitators to capture descriptions of promoting and hindering factors in delivering the intervention and data to optimize the training, research design and the protocol.
Replication and dissemination of the intervention | Baseline to 10 weeks
  Measured by an observational protocol of the intervention sessions, including (1) in-session behavior, (2) participant engagement, (3) social interaction within the group, (4) peer support and (5) change in perception of living with dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Ingelin Testad, PhD, Principal Investigator — Helse Stavanger HF
Locations (5):
- Neuroscience Research Australia, University of New South Wales, Sydney, New South Wales, Australia
- Norway (2):
  - Centre for Age-related Medicine (SESAM), Stavanger University Hospital, Stavanger, Rogaland
  - Norwegian National Advisory Unit on Ageing and Health, Oslo
- United Kingdom (2):
  - Cornwall Partnership NHS Foundation Trust, Bodmin, Cornwall
  - Devon Partnership NHS Trust, Exeter, Devon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Testad I, Clare L, Anstey K, Selbaek G, Bjorklof GH, Henderson C, Dalen I, Gjestsen MT, Rhodes S, Rosvik J, Bollen J, Amos J, Kajander MM, Quinn L, Knapp M. Self-management and HeAlth Promotion in Early-stage dementia with e-learning for carers (SHAPE): study protocol for a multi-centre randomised controlled trial. BMC Public Health. 2020 Oct 9;20(1):1508. doi: 10.1186/s12889-020-09590-9. PMID 33036591